CLINICAL TRIAL: NCT06484881
Title: Clinical Study of Probiotic Treatment for Androgenetic Alopecia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Concern about formulation patent
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Follea International Limited (Industry)
Responsible Party: Principal Investigator, Monica Naegle, Study Supervisor, Applied Biology, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA-001
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-06

CONDITIONS: Androgenetic Alopecia; Female Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Minoxidil 5% + Multivitamin Oral Supplement (Active Comparator): Topical Minoxidil 5% + Multivitamin Oral Supplement
  Interventions: Drug: Topical minoxidil 5%
- Placebo Spray + Daniel Alain Probiotic Treatment for Androgenetic Alopecia (Experimental): Placebo Spray + Daniel Alain Probiotic Treatment for Androgenetic Alopecia
  Interventions: Dietary Supplement: Daniel Alain Probiotic Treatment for Androgenetic Alopecia

INTERVENTIONS:
Dietary Supplement: Daniel Alain Probiotic Treatment for Androgenetic Alopecia — Probiotic
  Arms: Placebo Spray + Daniel Alain Probiotic Treatment for Androgenetic Alopecia
Drug: Topical minoxidil 5% — Topical minoxidil 5%
  Arms: Topical Minoxidil 5% + Multivitamin Oral Supplement

SUMMARY:
The primary objective of the study is to assess the efficacy of DA-001 as an oral supplement for treatment of female pattern hair loss.

DETAILED DESCRIPTION:
DA-001 is a botanical supplement demonstrated natural ingredients known to exert anti-androgen effects. The ingredients were tested in-vitro and have demonstrated the anti-androgen effect. This study aims to compare DA-001 to topical minoxidil in the treatment of female pattern hair loss (also known as androgenetic alopecia).

ELIGIBILITY:
Inclusion Criteria:

* Females Age 18 or older
* Diagnosed with female pattern hair loss
* Willing and able to apply the treatment as directed, comply with study
* Otherwise healthy
* Able to give informed consent

Exclusion Criteria:

* A medical history that may interfere with study objectives
* Women who are pregnant, lactating, or planning to become pregnant during the study period
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc)
* Subjects who have known allergies to any excipient in DA-001
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device in the treatment area within 30 days prior to study treatment initiation
* Subjects who have used any topical prescription medications in the treatment area within 30 days prior to study treatment initiation
* Subjects who have had a dermatological procedure such as surgery in the treatment area within 30 days prior to study treatment initiation
* Subject is unable to provide consent or make the allotted clinical visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects 18 and above
Enrollment: 0 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Target Area Hair Counts | Week [0,12]
  Target Area Hair Counts

CONTACTS AND LOCATIONS:
Overall Officials: Andy Goren, MD, Study Director — University of Rome G. Marconi

IPD SHARING:
Plan to Share IPD: No